CLINICAL TRIAL: NCT04963166
Title: Natural History of Systemic and Nasal Mucosal Immunity After Influenza Vaccination in a Pediatric Population
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000488; 000488-I
Record Dates: First submitted 2021-07-14; First posted 2021-07-15 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09-10

CONDITIONS: Influenza Immunity
Keywords: Flu; Flu Shot; Children; Natural History
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 12-17 years of age: 12-17 years of age
- 2-6 years of age: 2-6 years of age
- 7-11 years of age: 7-11 years of age

SUMMARY:
Background:

The influenza (flu) virus infects millions around the world every year. Children are at increased risk of complications from the flu. The flu vaccine protects against influenza, but the vaccine can be improved. Researchers want to learn more about children s mucosal and systemic immunity after flu vaccination. This could help to develop more effective flu vaccines in the future.

Objective:

To learn what happens in kids immune systems after receiving a flu vaccine.

Eligibility:

Children ages 2-17 who have received a flu vaccine in the past and plan to get the current seasonal flu vaccine given by injection.

Design:

All study visits will take place at home and communication with the study team will be done via phone or videoconference.

Participants will review medical history and flu vaccination history with the study team.

Participants will get the flu vaccine at their local doctor s office or pharmacy. They will not be given the vaccine in this study.

Participants will complete an electronic survey to give details about the date and type of flu vaccine received.

Participants will collect nasal and fingerstick samples at home. They will collect 4 nasal samples and 3 fingerstick samples over 6 months: once before they get the flu vaccine and 2-3 times after they get the vaccine. They will use collection kits that include instructions, sample collection supplies, and shipping materials. They will ship all samples back to NIH with all costs covered by NIH.

Participation will last for 6 months.

Compensation is provided.

DETAILED DESCRIPTION:
Title:

Natural History of Systemic and Nasal Mucosal Immunity after Influenza Vaccination in a Pediatric Population

Study Description:

While adults are heavily represented in influenza vaccine studies, there are limited studies in the pediatric population. This study will characterize the changes in nasal and systemic immunity after influenza vaccination in a pediatric population.

Objectives:

Primary Objectives:

Characterize nasal mucosal humoral immune response pre and post influenza vaccination

Characterize systemic humoral immune response pre and post influenza vaccination

Secondary Objectives:

Describe the trend of nasal mucosal mucosal and serum humoral immune response over time after vaccination

Endpoints:

Primary Endpoints:

1. Baseline and post-vaccination mucosal anti-influenza antibodies from nasal samples as measured by:

   1. Anti-hemagglutination (HA) head antibody quantitative enzyme-linked immunosorbent assay (ELISA) immunoglobulins (Ig) (IgA, IgG)
   2. Anti-HA stalk antibody quantitative ELISA (IgA, IgG)
   3. Anti-neuraminidase (NA) antibody quantitative ELISA (IgA, IgG)
2. Baseline and post-vaccination systemic anti-influenza antibodies as measured by:

   1. Anti-HA head antibody quantitative ELISA (IgM, IgG, IgA)
   2. Anti-HA stalk antibody quantitative ELISA (IgM, IgG, IgA)
   3. Anti-NA antibody quantitative ELISA (IgM, IgG, IgA)

Secondary Endpoints:

Multiple timepoint measurements of mucosal anti-influenza antibodies from nasal samples as measured by:

Anti-HA head antibody quantitative ELISA (IgA, IgG)

Anti-HA stalk antibody quantitative ELISA (IgA, IgG)

Anti-NA antibody quantitative ELISA (IgA, IgG)

Multiple timepoint measurements of systemic anti-influenza antibodies as measured by:

Anti-HA head antibody quantitative ELISA (IgM, IgG, IgA)

Anti-HA stalk antibody quantitative ELISA (IgM, IgG, IgA)

Anti-NA antibody quantitative ELISA (IgM, IgG, IgA)

Study Population:

Children who are >= 2 years and < 18 years of age (N = 51; accrual ceiling = 100). Participants will be enrolled by age group: 2 - 6 years old, 7 - 11 years old and 12 - 17 years old with a goal enrollment of 17 per group.

Description of Sites/Facilities Enrolling Participants:

Participants will be enrolled by telephone or videoconference, and sample collections will be done in participant homes. Recruitment will be from community pediatric clinics and self- or family referral.

Study Duration:

2 years

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to enroll in this study, an individual must meet all of the following criteria:

* >= 2 years of age and < 18 years of age at the time of enrollment.
* Completed a previous influenza series in the past and therefore requires only one seasonal influenza vaccine every year.
* Planning to receive the current seasonal inactivated influenza vaccine given by injection.
* Parent or guardian willing and able to provide verbal consent.
* Willing and able to undergo home blood micro-sampling and nasal sampling.
* Willing to have samples stored for future research.
* Parent/guardian able to proficiently speak, read, and write English.

EXCLUSION CRITERIA:

Any individual who meets any of the following criteria will be excluded from participation in this study:

* Already received the current season s influenza vaccine.
* Planning to receive the current seasonal live attenuated influenza vaccine (LAIV).
* Self-reported pregnancy or breastfeeding.
* Any condition that, in the opinion of the investigator, would compromise the safety of the study participant or staff, or would prevent proper conduct of the study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children receiving their first ever influenza vaccine require two doses of the vaccine one month apart and will not be included in this study. Only participants who have already received a flu vaccine series in the past will be eligible for this study. Evaluation of immunity after the first ever influenza vaccination series is an important question that should be explored separately. We will enroll participants into one of three cohorts by age: 2 6 years old, 7 11 years old, and 12 17 years old. We will aim to enroll similar numbers of participants into each group to ensure a diverse age range in our population.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Baseline and post-vaccination (6 weeks) systemic anti-influenza antibodies as measured by: 1. Anti-HA head antibody quantitative ELISA IgM, IgG, IgA 2. Anti-HA stalk antibody quantitative ELISA IgM, IgG, IgA 3. Anti-NA antibody quantitative ELIS... | 6 weeks
  Systemic anti-influenza antibodies
Baseline and post-vaccination (6 weeks) mucosal anti-influenza antibodies from nasal samples as measured by: 1. Anti-HA head antibody quantitative ELISA IgA, IgG 2. Anti-HA stalk antibody quantitative ELISA IgA IgG 3. Anti-NA antibody quantitati... | 6 weeks
  Mucosal anti-influenza antibodies

SECONDARY OUTCOMES:
post-vaccination systemic anti-influenza antibodies | 24 weeks
  Systemic anti-influenza antibodies
post-vaccination mucosal anti-influenza antibodies | 24 weeks
  Mucosal anti-influenza antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Alison Han, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
This is a small observational study, not an interventional trial, involving pediatric participants.